CLINICAL TRIAL: NCT04435483
Title: Phase I, Open-label, Single-dose, Sequential, Randomized, Crossover Study of Acalabrutinib Suspension Delivered Via Nasogastric Tube in Healthy Subjects to Evaluate Relative Bioavailability and Proton-pump Inhibitor (Rabeprazole) Effect
Brief Title: A Study of Acalabrutinib Suspension to Evaluate Relative Bioavailability and Proton-pump Inhibitor Effect in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Acerta Pharma, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D822FC00004
Record Dates: First submitted 2020-06-01; First posted 2020-06-17 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Pharmacokinetics; Bioavailability
Keywords: Calquence; Acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence 1 (Experimental): Participants will receive Treatment A (100 mg acalabrutinib suspension via NG administration plus 20 mg rabeprazole) in Period 1, Treatment B (100 mg acalabrutinib suspension via NG administration) in Period 2, and Treatment C (100 mg acalabrutinib capsule) in Period 3.
  Interventions: Drug: Acalabrutinib Treatment A; Drug: Acalabrutinib Treatment B; Drug: Acalabrutinib Treatment C
- Treatment Sequence 2 (Experimental): Participants will receive Treatment B (100 mg acalabrutinib suspension via NG administration) in Period 1, Treatment C (100 mg acalabrutinib capsule) in Period 2, and Treatment B (100 mg acalabrutinib suspension via NG administration) in Period 3.
  Interventions: Drug: Acalabrutinib Treatment B; Drug: Acalabrutinib Treatment C

INTERVENTIONS:
Drug: Acalabrutinib Treatment A — Participants will receive a single dose of 100-mg acalabrutinib suspension via NG administration, under fasted conditions. A single dose of 20 mg rabeprazole will be administered with 240 mL water, 2 hours prior to administration of acalabrutinib suspension. Treatment with rabeprazole 20 mg twice daily (with meals) will be started 3 days prior to the receiving the first dose of acalabrutinib suspension.
  Arms: Treatment Sequence 1
Drug: Acalabrutinib Treatment B — Participants will receive a single dose of 100-mg acalabrutinib suspension via NG administration, under fasted conditions.
Drug: Acalabrutinib Treatment C — Participants will receive a single dose of 100-mg acalabrutinib capsule, under fasted conditions. The acalabrutinib capsule will be administered with 240 mL of water.

SUMMARY:
This study is being conducted to support the clinical development of acalabrutinib in patients who are unable to swallow capsule and require nasogastric (NG) tube placement.

DETAILED DESCRIPTION:
This is an open-label, single-center, randomized, 3-period, crossover study of acalabrutinib suspension administered via NG tube in healthy subjects to evaluate the relative bioavailability and proton-pump inhibitor (rabeprazole) effect.

The study is divided in 3 periods.

Period 1 of the study is designed to investigate the effect of proton-pump inhibitor on the pharmacokinetics (PK) of acalabrutinib suspension. Period 2 and 3 of the study are designed to investigate the bioavailability of acalabrutinib suspension relative to an oral capsule formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study-specific procedures.
2. Healthy adult male and female subjects aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
3. Male subjects and their female partners/spouses must adhere to the contraception methods.
4. Female subjects must have a negative pregnancy test at screening, must not be lactating, and must be of non-childbearing potential.
5. Have a body mass index (BMI) between 18.5 and 30 kg/m2, inclusive, and weigh at least 50 kg and no more than 100 kg, inclusive, at screening.

Exclusion Criteria:

1. History or presence of any clinically significant disease (including COVID-19) or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History or presence of gastrointestinal (GI), hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any positive result on screening for serum hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
4. Plasma donation within 30 days of screening or any blood donation/loss more than 500 mL during the 90 days prior to screening.
5. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the 90 days prior to screening.
6. Positive screen for drugs of abuse or cotinine at screening.
7. Known or suspected history of alcohol or drug abuse, or excessive intake of alcohol as judged by the Investigator.
8. Excessive intake of caffeine-containing drinks or food as judged by the Investigator.
9. Vulnerable subjects, eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
10. History of a disorder which would make NG tube placement contraindicated, eg, esophageal strictures, esophageal varices, or bleeding diathesis.
11. Evidence of ongoing systemic bacterial, fungal, or viral infection (including upper respiratory tract infections). Subjects with localized cutaneous fungal infections are eligible.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Acalabrutinib and ACP-5862 plasma PK parameter: Area under plasma concentration-time curve from time zero to infinity (AUCinf) | Day 1 to 2: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours (h) post-dose
  To compare the AUCinf of the acala NG suspension with and without rabeprazole. To compare the AUC of the acala NG suspension with the oral capsule.
Acalabrutinib and ACP-5862 plasma PK parameter: Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUClast) | Day 1 to 2: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h post-dose
  To compare the AUClast of the acala NG suspension with and without rabeprazole. To compare the AUClast of the acala NG suspension with the oral capsule.
Acalabrutinib and ACP-5862 plasma PK parameter: Maximum observed plasma concentration (Cmax) | Day 1 to 2: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h post-dose
  To compare the Cmax of the acala NG suspension with and without rabeprazole. To compare the Cmax of the acala NG suspension with the oral capsule.

SECONDARY OUTCOMES:
Acalabrutinib and ACP-5862 plasma PK parameter: Area under the plasma concentration-time curve from time zero to 24 hours post-dose (AUC0-24) | Day 1 to 2: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h post-dose
  To compare the AUC0-24 of the acala NG suspension with and without rabeprazole. To compare the AUC0-24 of the acala NG suspension with the oral capsule.
Acalabrutinib and ACP-5862 plasma PK parameter: Time to reach maximum observed plasma concentration (tmax) | Day 1 to 2: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h post-dose
  To compare the tmax of the acala NG suspension with and without rabeprazole. To compare the tmax of the acala NG suspension with the oral capsule.
Acalabrutinib and ACP-5862 plasma PK parameter: Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t1/2) | Day 1 to 2: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h post-dose
  To compare the t1/2 of the acala NG suspension with and without rabeprazole. To compare the t1/2 of the acala NG suspension with the oral capsule.
Acalabrutinib and ACP-5862 plasma PK parameter: Mean residence time of the drug in the systemic circulation from zero to infinity (MRT) | Day 1 to 2: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h post-dose
  To compare the MRT of the acala NG suspension with and without rabeprazole. To compare the MRT of the acala NG suspension with the oral capsule.
Acalabrutinib and ACP-5862 plasma PK parameter: Terminal elimination rate constant (λz) | Day 1 to 2: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h post-dose
  To compare the λz of the acala NG suspension with and without rabeprazole. To compare the λz of the acala NG suspension with the oral capsule.
Acalabrutinib and ACP-5862 plasma PK parameter: Apparent total body clearance of drug from plasma after extravascular administration (acalabrutinib only) (CL/F) | Day 1 to 2: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h post-dose
  To compare the CL/F of the acala NG suspension with and without rabeprazole. To compare the CL/F of the acala NG suspension with the oral capsule.
Acalabrutinib and ACP-5862 plasma PK parameter: Apparent volume of distribution during the terminal phase after extravascular administration (acalabrutinib only) (Vz/F) | Day 1 to 2: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h post-dose
  To compare the Vz/F of the acala NG suspension with and without rabeprazole. To compare the Vz/F of the acala NG suspension with the oral capsule.
Acalabrutinib and ACP-5862 plasma PK parameter: Metabolite to parent ratio based on AUCinf and/or AUClast (M:P[AUC]) | Day 1 to 2: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h post-dose
  To compare the M:P[AUC] of the acala NG suspension with and without rabeprazole. To compare the M:P[AUC] of the acala NG suspension with the oral capsule.
Acalabrutinib and ACP-5862 plasma PK parameter: Metabolite to parent ratio based on Cmax (M:P[Cmax]) | Day 1 to 2: Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24 h post-dose
  To compare the M:P[Cmax] of the acala NG suspension with and without rabeprazole. To compare the M:P[Cmax] of the acala NG suspension with the oral capsule.
Number of subjects with abnormal vital signs | Screening, Day -1, and Day 2
  To assess the safety and tolerability of single doses of acalabrutinib suspension in healthy participants.
Number of subjects with abnormal laboratory assessments | Screening, Day -1, Days 1-2, and follow-up visit (7-10 days after last dose)
  To assess the safety and tolerability of single doses of acalabrutinib suspension in healthy participants.
Number of subjects with serious and non-serious adverse events | Screening (Day -28), Days -3, -2, -1, Days 1-3, and follow-up visit (7-10 days after last dose)
  To assess the safety and tolerability of single doses of acalabrutinib suspension in healthy participants.

CONTACTS AND LOCATIONS:
Overall Officials: David Han, M.D., Principal Investigator — PAREXEL Early Phase Clinical Unit-Los Angeles
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home